CLINICAL TRIAL: NCT04483622
Title: Immunoglobulin G Antibody Immune Response Profile Following Infection With SARS-CoV-2 in COVID-19 Egyptian Patients
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Goda, assistant professor of medical microbiology and immunology at sohag faculty of medicine fa, Sohag University
Other Study IDs: IBR#S20-133
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Covid19
Keywords: COVID19 IGg
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to detect the evidence on the immune response following acute SARS-CoV-2 infections. the study will report the profile of IgG specific antibodies levels to SARS-CoV-2 infection found in recovered coronavirus disease (COVID-19) patients after infection for both symptomatic and asymptomatic patients.

DETAILED DESCRIPTION:
A total of 30 COVID-19 patients for the study will be enrolled. All the patients enrolled were confirmed to be infected with SARS-CoV-2 by RT-PCR assay for nasal and pharyngeal swab specimens.

For the study, serum samples of the 30 patients will be collected and will be investigated for the detection rate for immunoglobulin G (IgG). The first sample will be collected 2 weeks after the second negative RT-PCR assay for nasal and pharyngeal swab specimens and 6 samples will be collected after that for 6 months later; one serum sample tested every month for 6 months after.

The following questions will be addressed:-

1. What proportion of confirmed cases develops specific IgG antibodies to SARS-CoV-2?
2. How long is the duration of detection of serum IgG antibodies and antibody titres over time following infection with SARS-CoV-2?

ELIGIBILITY:
Inclusion Criteria:

* patients with recent COVID- 19 infection(2 weeks after the second negative RT-PCR assay)

Exclusion Criteria:

* patients on immune-suppressive therapy
* patients with immunological disease

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients attending sohag university hospital and have recent COVID -19 infection
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
rising titre of IGg antibodies | first month
  it's expected to have COVID-19 antibodies within 1month of infection the antibody titre expected to rise the fall to a lower levels

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No